CLINICAL TRIAL: NCT05512689
Title: Optimization of Ventilation Strategies in Preterm and Term Infants in a Single-center Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Michael Wagner, Principal Investigator, Medical University of Vienna
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 1334/2022
Record Dates: First submitted 2022-08-18; First posted 2022-08-23 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Lung-protective Ventilation; Respiratory Function Monitor

STUDY DESIGN:
Intervention Model Description: We aimed to avoid classical randomization due to a possible learning and habituation effect from the feedback when using the RFM. We started with a phase of routine ventilation, in which the healthcare professional ventilated the infants using the RFM but did not receive any feedback about the ventilation. This represents the normal clinical setting. In the second phase, the healthcare professional then received visual feedback from the RFM during ventilations. The healthcare professional could then adjust his ventilation technique in real time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): In the control group, the healthcare professional ventilates the infants without any feedback about the ventilation. This represents the normal clinical setting. The RFM will be recording data on the ventilation quality.
- Interventional group (Active Comparator): In the interventional group, healthcare professionals will ventilate the infants using the RFM and are able to adapt their ventilations according to the RFM feedback.
  Interventions: Device: Ventilations while using a respiratory function monitor

INTERVENTIONS:
Device: Ventilations while using a respiratory function monitor — Healthcare professionals are able to use a feedback device to guide their ventilations.
  Arms: Interventional group

SUMMARY:
This study was a non-blinded, non-randomized intervention study in a single-center clinical setting, analyzing ventilation quality with and without RFM visibility.

DETAILED DESCRIPTION:
The study was conducted at the Neonatal Intensive Care Unit and the delivery room at the Division of Neonatology, at the Medical University of Vienna.

We aimed to record ventilation parameters (tidal volume, mask leak, ventilation rate, PIP, PEEP) using a CE-certified Respiratory Function Monitor (Neo100, Monivent AB, Gothenburg, Sweden), which was either hidden or visible to the provider responsible for the airway (airway provider), during ventilations on term and preterm patients at the NICU and the delivery room.

The investigators aimed to determine the quality of ventilations performed by healthcare professionals depending on RFM visibility. Analysis occurred, determining whether observing the data displayed on the RFM during PPV of preterm and newborn infants lead to adjustments in applied pressure and an increase in the proportion of inflations performed within a predefined range of 4-8 ml/kg for VTe.

The investigators hypothesized that using a RFM with numeric and graphical display of values during positive pressure ventilation of infants will lead to i) more frequent recognition and correction of tidal volumes outside the predefined range and ii) reduction of mask leak.

This knowledge gain may improve future training using a RFM to improve the quality of ventilations and, thereby, patient safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients at the Neonatal Intensive Care Unit (NICU) and in the delivery room who receive positive pressure ventilation
* Written consent from parents or legal guardians of patients
* Preterm and term infants (male and female, any gestational age)

Exclusion Criteria:

- Healthcare professionals or parents/legal guardians, representing their children, that do not consent to participation in this study

Max Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Proportion of ventilations with VTe between 4-8ml/kg | through study completion, an average of 1 year
  percentage of ventilations within range divided through all ventilations performed, for each participant

SECONDARY OUTCOMES:
Mean value for mask leak and proportion of ventilations with excessive mask leak (defined as >50%) during all ventilations | through study completion, an average of 1 year
  defined as > 50%
Occurrence of insufficient tidal volume (defined as <4mL/kg) as a proportion of ventilations given (face mask and endotracheal tube) | through study completion, an average of 1 year
  defined as < 4ml/kg
Occurrence of excessive tidal volume (defined as >8mL/kg) as a proportion of ventilations given (face mask and endotracheal tube) | through study completion, an average of 1 year
  defined as > 8ml/kg
Mean value for ventilation rate (defined as ventilations per minute) | through study completion, an average of 1 year
  defined as ventilations per minute
Mean value for peak inflation pressure | through study completion, an average of 1 year
  defined as > 35 cmH2O
Outcome data and adverse events | through study completion, an average of 1 year
  this included diagnoses (i.e., bronchopulmonary dysplasia [BPD], persistent ductus arteriosus [PDA], IVH, periventricular leukomalacia [PVL], and pneumothorax) and the time frame of occurrence (within 24 hours, one week, or during the total hospital stay). BPD was defined as the need of any respiratory support at the GA of 36 weeks, evaluated for infants below 32+0 weeks GA. IVH was determined using the DEGUM classification
Comparison of elective versus delivery room interventions | through study completion, an average of 1 year
  mean values for all evaluated ventilation parameters (VTe, leak, PIP, rate) for this comparison
Comparison of fellows vs. consultants | through study completion, an average of 1 year
  mean values for all evaluated ventilation parameters (VTe, leak, PIP, rate) for this comparison
Comparison of sef-inflating-bag vs. neo-T | through study completion, an average of 1 year
  mean values for all evaluated ventilation parameters (VTe, leak, PIP, rate) for this comparison
Comparison of ventilations via face mask vs. endotracheal tube | through study completion, an average of 1 year
  mean values for all evaluated ventilation parameters (VTe, leak, PIP, rate) for this comparison

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wagner, MD PhD, Study Director — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
IPD will not be made available to other researchers.